CLINICAL TRIAL: NCT02617966
Title: Rod and Cone Mediated Function in Retinal Disease
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160024; 16-EI-0024
Record Dates: First submitted 2015-11-28; First posted 2015-12-01 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-08-12

CONDITIONS: Retinal Degeneration; Retinitis Pigmentosa; Stargardt's Disease
Keywords: Retina; Retinal Degeneration; Retinitis Pigmentosa; Stargardt's Disease; Dark Adaptation
MeSH Terms: conditions — Retinal Degeneration; Retinitis Pigmentosa; Stargardt Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Participants with retinal disease
- Unaffected: Healthy volunteers

SUMMARY:
Background:

Retinal diseases cause the loss of rod and cone photoreceptors. Symptoms include vision loss and night blindness. Researchers want to learn about rod and cone function in healthy people and people with retinal disease. They want to know if how well a person sees in the dark can test the severity of retinal disease.

Objectives:

To find out if how well a person sees in the dark can test the severity of retinal disease. To find out if this can help detect retinal disease and track its changes.

Eligibility:

People ages 5 and older with:

Retinal disease OR

20/20 vision or better with or without correction in at least one eye

Design:

Participants will be screened with medical and eye history and eye exam. Those with retinal disease will also have:

Eye imaging: Drops dilate the eye and pictures are taken of it.

Visual field testing: Participants look into a bowl and press a button when they see light.

Electroretinogram (ERG): An electrode is taped to the forehead. Participants sit in the

dark with their eyes patched for 30 minutes. Then they get numbing drops and contact

lenses. Participants watch lights while retina signals are recorded.

Visit 1 will be 3-8 hours. Participants will have up to 6 more visits over 6-12 months. Visits include:

Eye exam and imaging

Time course of dark adaptation: Participants view a background light for 5 minutes then

push a button when they see colored light.

Dark adapted sensitivity: Participants sit in the dark for 45 minutes. They push a button when

they see colored light.

For participants with retinal disease, ERG and visual field testing

...

DETAILED DESCRIPTION:
Objective: The objective of this protocol is to investigate local changes in rod and cone photoreceptor function across the retina in healthy volunteers and participants with retinal disease.

Study Population: Up to 250 healthy volunteers and 250 participants, age five or older, with retinal disease.

Design: This single-center, observational, case-control study will be comprised of three related Aims that assess rod and cone function with commercial perimeters and/or a commercial Cambridge Research Systems computer monitor (Display++) specialized for displaying stimuli at low light intensities. For Aim 1 the normal retinal sensitivity ranges will be established for both fundus-guided and non-guided perimeters. For Aim 2, the normal range for describing the kinetics of dark adaptation following bleaching of retinal rhodopsin will be established for the fundus-guided and non-guided perimeters. For Aim 3, local changes in rod and cone photoreceptor function across the retina in participants with retinal disease will be examined from measurement of the kinetics of dark adaptation, scotopic and photopic retinal sensitivity, and/or Radial Frequency (RF) hyperacuity on the Display++ monitor. Testing may also include patient reported outcome (PRO) questionnaires to assess vision problems under low luminance conditions.

Outcome Measures: The primary outcome for this study is to establish normal ranges for A) the kinetics of dark adaptation (time), B) retinal sensitivity (dB) for the fundus-guided and non-guided perimeters, and C) RF hyperacuity on the Display++ monitor. The secondary outcomes will be to examine changes in the kinetics of dark adaptation, scotopic and photopic retinal sensitivity, and/or RF hyperacuity in participants with retinal disease and potentially correlate these clinical measures with patients self-reported evaluation of their vision under low luminance conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant must be five years of age or older.
* Participant (or legal guardian) must understand and sign the protocol s informed consent document.
* Participant must be able to cooperate with the testing required for this study.

For Participants with retinal disease only:

* Participant must have retinal disease, defined as evidence of loss of retinal dysfunction and/or degeneration as established by standard clinical methods including perimetry, ERG and imaging.
* Participant must have a measurable visual acuity.

For Healthy Volunteers only:

-Participant must have visual acuity of 20/20 or better, with or without correction (e.g., glasses or contact lens) in at least one eye.

EXCLUSION CRITERIA:

-Participant with changes in pre-retinal media sufficient to obscure a view of the retina.

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 250 participants with retinal disease will be enrolled and up to 120 healthy volunteers will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes for this study are to establish normal ranges for the kinetics of dark adaptation and dark-adapted retinal sensitivity for the fundus guided and non-guided perimeters and for RF hyperacuity on the Display++. | ongoing, up to 10 visits in 5 years
  The primary outcomes for this study are to establish normal ranges for the kinetics of dark adaptation and dark-adapted retinal sensitivity for the fundus guided and non-guided perimeters and for RF hyperacuity on the Display++.

SECONDARY OUTCOMES:
Secondary outcomes will be to examine changes in the kinetics of dark adaptation and dark-adapted retinal sensitivity, and scotopic and photopic RF hyperacuity in participants with retinal disease. | ongoing, up to four visits in 5 years
  Secondary outcomes will be to examine changes in the kinetics of dark adaptation and dark-adapted retinal sensitivity, and scotopic and photopic RF hyperacuity in participants with retinal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Brett G Jeffrey, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jackson GR, Owsley C, Curcio CA. Photoreceptor degeneration and dysfunction in aging and age-related maculopathy. Ageing Res Rev. 2002 Jun;1(3):381-96. doi: 10.1016/s1568-1637(02)00007-7. PMID 12067593
- [Background] Massof RW, Finkelstein D. Rod sensitivity relative to cone sensitivity in retinitis pigmentosa. Invest Ophthalmol Vis Sci. 1979 Mar;18(3):263-72. PMID 422332
- [Background] Birch DG, Wen Y, Locke K, Hood DC. Rod sensitivity, cone sensitivity, and photoreceptor layer thickness in retinal degenerative diseases. Invest Ophthalmol Vis Sci. 2011 Sep 9;52(10):7141-7. doi: 10.1167/iovs.11-7509. PMID 21810977
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-EI-0024.html